CLINICAL TRIAL: NCT07365449
Title: Visual Versus Conventional Intubation: Comparison of SaCoVLM™ Video Laryngeal Mask and Direct Laryngoscopy : A Prospective Observational Study
Brief Title: Visual Versus Conventional Intubation Using the SaCoVLM Video Laryngeal Mask
Acronym: SACOV-VS-DL
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Emel Gunduz, Associate Professor of Anesthesiology, Akdeniz University, Antalya, Turkey, Akdeniz University
Other Study IDs: AKDENIZ_SACOVLM_INTUBATION_01
Record Dates: First submitted 2025-11-26; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Airway Management
Keywords: Airway management;; Video laryngoscopy;; Hemodynamics;; Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: SaCoVLM™ Video Laryngeal Mask Group 2: Direct Laryngoscopy: Group 1: SaCoVLM™ Video Laryngeal Mask (VLM), "Intubation performed using SaCoVLM™ video laryngeal mask under general anesthesia."
  Group 2: Direct Laryngoscopy (DL),: "Intubation performed using direct laryngoscopy under general anesthesia."

SUMMARY:
This is a prospective, observational study designed to evaluate airway management techniques used during elective surgery under general anesthesia. The study focuses on perioperative hemodynamic parameters and airway-related procedural characteristics.

DETAILED DESCRIPTION:
Study Design This is a single-center, prospective, observational study conducted at Akdeniz University Hospital after approval by the Institutional Ethics Committee (Approval No: 70904504/139). Written informed consent was obtained from all participants prior to enrollment.

Participants Adult patients scheduled for elective surgery under general anesthesia between March and June 2024 were screened for inclusion.

Exclusion Criteria Patients were excluded if they were under 18 years of age, pregnant, had known hypersensitivity to anesthetic agents, gastroesophageal reflux disease, or active upper respiratory tract infection.

Group Allocation and Airway Management

Due to the observational design of the study, randomization was not performed. Patients were allocated to groups according to the airway management technique selected by the attending anesthesiologist:

SaCoVLM™ video laryngeal mask group (VLM)

Direct laryngoscopy group (DL)

All airway procedures were performed by anesthesiologists with at least three years of clinical experience and a minimum of 50 prior successful supraglottic airway device and endotracheal intubations.

Devices The SaCoVLM™ is a video-integrated supraglottic airway device with separate channels for ventilation, visualization, and gastric access. Mask size selection was based on patient body weight.

In the DL group, Macintosh laryngoscope blades (sizes 3 or 4) were used according to clinician preference.

Preoperative Assessment Pre-induction airway evaluation included Mallampati score, upper lip bite test, neck circumference, thyromental distance, sternomental distance, and interincisor gap. The STOP-Bang questionnaire was completed preoperatively.

Anesthesia Protocol All patients fasted for at least 8 hours for solids and 6 hours for liquids. Standard monitoring included ECG, non-invasive blood pressure, pulse oximetry, bispectral index (BIS), and capnography.

Preoxygenation was performed with 80% oxygen for 2 minutes. Anesthesia induction was achieved using thiopental, fentanyl, lidocaine, and rocuronium. Airway intervention was initiated once BIS values decreased below 50.

Airway Procedure and Measurements In the VLM group, the time from device insertion to visualization of the glottis was recorded. After confirmation of ventilation using capnography, a lubricated endotracheal tube was advanced through the device, and the time from tube insertion to passage through the vocal cords was recorded.

In the DL group, the time from laryngoscope insertion to passage of the endotracheal tube through the vocal cords was recorded.

Glottic visualization was assessed using the SaCoVLM™ visualization scale in the VLM group and the Cormack-Lehane classification in the DL group.

Cuff pressures were maintained below 60 cmH₂O for the laryngeal mask and below 25 cmH₂O for endotracheal tubes.

Hemodynamic Monitoring Hemodynamic parameters including systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate, and oxygen saturation were recorded at predefined time points: preoperative baseline, post-induction, post-laryngeal mask insertion, and post-endotracheal tube placement.

Maintenance and Emergence Anesthesia was maintained with sevoflurane titrated to a BIS value of 40-60 and a remifentanil infusion. At the end of surgery, anesthetic agents were discontinued and extubation was performed once patients regained consciousness and responded to verbal commands.

Outcome Measures Primary outcomes included hemodynamic responses to airway management, first-attempt success, airway procedure time, and airway-related complications.

Secondary outcomes included the need for adjunct airway maneuvers, glottic visualization grading, and postoperative airway-related adverse events.

Sample Size Calculation Sample size estimation was based on prior literature using an effect size of 1.68, an alpha level of 0.05, and a statistical power of 95%, resulting in a minimum required sample size of 22 patients per group.

Statistical Analysis Statistical analysis was planned using appropriate parametric methods following assessment of data distribution. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Scheduled for elective surgery under general anesthesia

Requires tracheal intubation as part of the planned anesthetic technique

American Society of Anesthesiologists (ASA) physical status I-III

Able to provide written informed consent

Exclusion Criteria:

Age < 18 years

Pregnancy

Known or suspected hypersensitivity to anesthetic agents used in the protocol

History of gastroesophageal reflux disease or increased risk of aspiration

Active upper respiratory tract infection

Predicted difficult airway (Mallampati class IV, mouth opening < 3 cm, limited neck mobility)

Severe cardiopulmonary instability

Emergency surgery

Upper airway pathology (airway trauma, tumor, edema, infection)

Coagulopathy or bleeding tendency

Inability to cooperate or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included adult patients (≥18 years old) scheduled for elective surgery under general anesthesia at Akdeniz University Hospital between March and June 2024. Both male and female patients were eligible. Patients with known hypersensitivity to anesthetic agents, pregnant patients, those with gastroesophageal reflux disease, or active upper respiratory tract infections were excluded. A total of 204 patients were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Mean Arterial Pressure During Intubation | Baseline (pre-induction) and 1 minute after endotracheal tube placement
  Mean arterial pressure (MAP) measured non-invasively at baseline (before induction of anesthesia) and at 1 minute after successful endotracheal tube placement.

SECONDARY OUTCOMES:
First-Attempt Intubation Success | During airway instrumentation (peri-procedural) Unit of Measure Percentage (%)
  Successful placement of the endotracheal tube on the first attempt, confirmed by continuous capnography.
Heart Rate Response to Intubation | Baseline (pre-induction) and 1 minute after endotracheal tube placement Unit of Measure beats per minute
  Heart rate measured at baseline (before induction of anesthesia) and at 1 minute after endotracheal tube placement.
Oxygen Saturation During Airway Management | Baseline and during airway instrumentation Unit of Measure Percentage (%)
  Peripheral oxygen saturation (SpO₂) measured at baseline and during airway instrumentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Please Select:, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared with other researchers

REFERENCES:
- [Result] Yan CL, Chen Y, Sun P, Qv ZY, Zuo MZ. Preliminary evaluation of SaCoVLM video laryngeal mask airway in airway management for general anesthesia. BMC Anesthesiol. 2022 Jan 3;22(1):3. doi: 10.1186/s12871-021-01541-0. PMID 34979936
- [Result] Yan CL, Zhang YQ, Chen Y, Qv ZY, Zuo MZ. To compare the influence of blind insertion and up-down optimized glottic exposure manoeuvre on oropharyngeal leak pressure using SaCoVLM video laryngeal mask among patients undergoing general anesthesia. J Clin Monit Comput. 2023 Apr;37(2):593-598. doi: 10.1007/s10877-022-00930-1. Epub 2022 Oct 29. PMID 36308611